CLINICAL TRIAL: NCT07360028
Title: Efficacy of Ultrasound Guided Erector Spinae Plane Block Versus Ultrasound Guided Serratus Anterior Plane Block for Postoperative Pain Control Following Video-assisted Thoracoscopic Surgeries (VATS): Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD 307/2025
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain Control
Keywords: post operative pain control
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erectror Spinae Plane Block (Active Comparator): Ultrasound Guided block using 20 mL of 0.25% bupivacaine.
  Interventions: Procedure: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®)
- Serratus Anterior Plane Block (Active Comparator): Ultrasound Guided block using 20 mL of 0.25% bupivacaine.
  Interventions: Procedure: Serratus anterior plane block (SAP)

INTERVENTIONS:
Procedure: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) — Ultrasound Guided Erector Spinae Plane block using 20 mL of 0.25% bupivacaine.
  Arms: Erectror Spinae Plane Block
Procedure: Serratus anterior plane block (SAP) — Ultrasound Guided Serratus Anterior Plane Block using 20 mL of 0.25% bupivacaine.
  Arms: Serratus Anterior Plane Block

SUMMARY:
The aim of the study is to compare the analgesic efficacy of Erector spinae plane block versus Serratus anterior plane block in patients undergoing video-assisted thoracoscopic surgeries.

DETAILED DESCRIPTION:
The aim of the study is to compare the analgesic efficacy of Erector spinae plane block versus Serratus anterior plane block in patients undergoing video-assisted thoracoscopic surgeries.

Preoperative: - On the day before surgery, all patients will be evaluated, detailed medical and surgical history will be taken also physical and systemic examinations will be done.

The following investigations will be done including complete blood count, liver enzymes, prothrombin time, partial thromboplastin time, International normalized ratio (INR) , kidney functions, serum electrolytes and ECG.

All patients will be informed about the visual analogue scale (VAS) on a scale from 0 to 10 where 0 represents no pain and 10 represents the worst imaginable pain.

In the pre-Anesthetic room:

* baseline hemodynamics will be recorded including heart rate (HR) and mean arterial blood pressure (MAP) and An intravenous access will be inserted.
* In the operating theatre, full monitors will be applied. Intraoperative: -
* Fentanyl (1 μg/kg), propofol (2 mg/kg) and atracurium(0.5 mg/kg) will be given IV for general anesthesia induction.
* Intubation will be done using a double-lumen endobronchial tube size 37 Fr in females and 39 Fr in males, tidal volume will be 6-8 ml/kg in case of both lungs ventilation and 4-6ml/kg during singe lung ventilation.

Anesthesia will continue using isoflurane 2 vol. %, 50% O2 and 50% air.

* Moreover, three milligrams of Granisetron will be given as prophylactic against nausea and vomiting post-operatively.
* During operation, 6 mL/kg/h of Ringer's solution will be administered.
* At the end of surgery, the patient will be positioned laterally.
* All blocks will be done using ultrasound-guidance (Mindray ultrasound) using high frequency linear probe (10-12 MHZ) by the same experienced senior doctors.

Group A : (25 patients) patients will receive Erector Spinae Plane Block using 20 mL of 0.25% bupivacaine.

Group B: (25 patients) patients will recieve Serratus Aneterior Plane Block using 20 mL of 0.25% bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiology physical status ASA I, II and III.
* Patients aged between 25 and 70 years.
* patients undergoing video-assisted thoracoscopic surgeries (VATS), including pleurectomy, bullectomy, sympathectomy, esophagectomy, decortication, lobectomy, and pneumonectomy.

Exclusion Criteria:

* Patients below age of 25 or above age of 70.
* Patient refusal.
* Allergy to local anesthetic drugs.
* Bleeding or coagulation disorder.
* Psychiatric disorders.
* Infection at the needle entry site.
* Renal impairment (creatinine >1.5 ).
* Hepatic impairment (Child B or C).
* Patients with known Cortisol related diseases such as Cushing's Syndrome or Addison's Disease.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for Assessing postoperative pain control | after ICU admission at 2, 4, 8, 16, 24 hours post operative.
  Assessing The difference in postoperative pain control between both groups as determined by assessing the visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Abbassia-Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No